CLINICAL TRIAL: NCT00812500
Title: Dietary Protein Requirement of Elderly Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Prof. Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00-226
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2008-12

CONDITIONS: Age
Keywords: assess the effect of age on the EAR and RDA for protein

ARMS (4):
- 1 (Experimental): Young men, age 21-46 years.
  Interventions: Other: Lower Protein; Other: Medium Protein; Other: Higher Protein
- 2 (Experimental): Old Men, age 63-81 years.
  Interventions: Other: Lower Protein; Other: Medium Protein; Other: Higher Protein
- 3 (Experimental): Young women, age 21-46 years.
  Interventions: Other: Lower Protein; Other: Medium Protein; Other: Higher Protein
- 4 (Experimental): Old women, age 63-81 years.
  Interventions: Other: Lower Protein; Other: Medium Protein; Other: Higher Protein

INTERVENTIONS:
Other: Lower Protein — Each subject completed an 18-day periods (trials) of strict dietary control of consuming a lower protein diet.
Other: Medium Protein — Each subject completed an 18-day periods (trials) of strict dietary control of consuming a medium protein diet.
Other: Higher Protein — Each subject completed an 18-day periods (trials) of strict dietary control of consuming a higher protein diet.

SUMMARY:
The purpose of this study was to assess the effect of age on the estimated average requirement and adequate allowance for dietary protein.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-46 years, 63-81 years old
* Not diagnosed with diabetes or metabolic syndrome
* Clinically normal blood laboratory values

Exclusion Criteria:

* Age: 21 years of younger, 47-62 years old, and 82 years and older
* BMI: 20-29 kg/m
* Weight stable: <2kg change within the last 3 months
* Physical Activity: constant habitual pattern, no deviation >1x week of 30/minute sessions within the last 3 months

Clinically abnormal values:

* Blood
* Urine

Also, exclude any:

* Using meds that would influence appetite
* Using any anti-inflammatory steroid medications
* Has a joint replacement
* A medical condition that might place them at risk for participating in the study or interfere with successful completion of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-05; Primary Completion 2003-05 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To determine the dietary protein requirement of older men and women. | 57 days

SECONDARY OUTCOMES:
What is the lowest amount of protein that a man or women should eat each day to help him or her stay healthy? | 57 days

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States